CLINICAL TRIAL: NCT04924530
Title: Revealing the Mechanisms by Which Milk Sugars Exaggerate Postprandial Lipaemia
Brief Title: Effect of Lactose on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Oxford (Other); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19/NW/0630
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Risk Factor; Lipaemia; Metabolic Disease
MeSH Terms: conditions — Hyperlipidemias; Metabolic Diseases | interventions — maltodextrin; Sucrose; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maltodextrin (Sham Comparator): Glucose polymer; a common sugar substitute
  Interventions: Dietary Supplement: Maltodextrin
- Sucrose (Active Comparator): Fructose-glucose disaccharide
  Interventions: Dietary Supplement: Sucrose
- Lactose (Experimental): Galactose-glucose disaccharide
  Interventions: Dietary Supplement: Lactose

INTERVENTIONS:
Dietary Supplement: Maltodextrin — Co-ingestion of maltodextrin with a high fat meal
  Arms: Maltodextrin
Dietary Supplement: Sucrose — Co-ingestion of sucrose with a high fat meal
  Arms: Sucrose
Dietary Supplement: Lactose — Co-ingestion of lactose with a high fat meal
  Arms: Lactose

SUMMARY:
This study aims to determine to what extent ingestion of free sugars influence postprandial triglyceridaemia in men and women.

DETAILED DESCRIPTION:
Each participant will undergo three experimental trials in a randomized, crossover research design. On each study day, participants will consume a test drink containing standardised amounts of carbohydrate and fat followed by collection of blood and breath samples to assess metabolic responses during the 6 hour postprandial period. Trials will be identical except for the type of carbohydrate contained within the test drink: 1) maltodextrin (glucose polymer), 2) lactose (galactose-glucose disaccharide) and 3) sucrose (fructose-glucose disaccharide).

ELIGIBILITY:
Inclusion Criteria:

• Age: 18-50 years and premenopausal (for women)

Exclusion criteria:

* Weight instability (>5 kg change in body mass within last 6 months)
* Diagnosis of any form of diabetes
* Intolerances or allergies to any of the study procedures (e.g. lactose intolerance)
* Galactose disorders (e.g. galactokinase deficiency, UDPgalactose-4-epimerase deficiency, galactose-1-phosphate uridyl transferase deficiency)
* Fructose malabsorption
* Inborn errors of fructose metabolism (e.g. fructokinase deficiency, aldolase B deficiency, fructose-1,6-bisphosphatase deficiency)
* Pregnant or lactating
* Any condition that could introduce bias to the study (e.g. diagnoses of lipid disorders, including cardiovascular disease, or therapies that alter lipid or glucose metabolism, such as statins or niacin).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Raw data will be made available online upon publication in a peer-reviewed journal.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 dropouts
Groups:
- Sequence 1: Sucrose first, then Lactose, then Maltodextrin
- Sequence 2: Sucrose first, then Maltodextrin, then Lactose
- Sequence 3: Lactose first, then Sucrose, then Maltodextrin
- Sequence 4: Lactose first, then Maltodextrin, then Sucrose
- Sequence 5: Maltodextrin first, then Sucrose, then Lactose
- Sequence 6: Maltodextrin first, then Lactose, then Sucrose
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 3 | 4 | 2 | 4 | 4
Completed | 7 (Crossover design so n = 24 for the total n and for each arm.) | 3 (Crossover design so n = 24 for the total n and for each arm.) | 4 (Crossover design so n = 24 for the total n and for each arm.) | 2 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 3 | 4 | 2 | 4 | 4
Completed | 7 | 3 | 4 | 2 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 3 | 4 | 2 | 4 | 4
Completed | 7 | 3 | 4 | 2 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Crossover design so n = 24 for all arms
Groups:
- All Study Participants: All participants completed all conditions/arms and hence are pooled for baseline measures
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24
Height (m) [Mean (Standard Deviation); unit: meters] | 1.77 (0.11)
Body mass (kg) [Mean (Standard Deviation); unit: kg] | 72.7 (12.9)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] | 23.3 (2.2)
Body fat (percentage of mass) [Mean (Standard Deviation); unit: %] | 27 (9)
Fat mass (kg) [Mean (Standard Deviation); unit: kg] | 19.4 (7.3)
Fat-free mass (kg) [Mean (Standard Deviation); unit: kg] | 53.8 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Changes in Plasma Triglyceride Concentrations
Description: Incremental area under the curve (iAUC) of plasma triglyceride concentrations from timepoints 0, 30, 60, 120, 180, 240, 300, 360 minutes
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mmol/L x 360 min
Arm/Group | Maltodextrin | Sucrose | Lactose
Number analyzed (Participants) | 24 | 24 | 24
mmol/L x 360 min | 51 (68) | 90 (95) | 98 (88)

2. Secondary Outcome: Postprandial de Novo Lipogenesis (DNL)
Description: Time course for synthesis of fatty acids from non-lipid precursors using stable isotope methodology
Time Frame: 6 hours
Reporting Status: Not Posted

3. Secondary Outcome: Dietary Fat Oxidation
Description: Time course for whole-body dietary fatty acid oxidation using stable isotope methodology
Time Frame: 6 hours
Reporting Status: Not Posted

4. Secondary Outcome: Postprandial Changes in Plasma Insulin Concentrations
Description: Incremental area under the curve (iAUC) of plasma insulin concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

5. Secondary Outcome: Postprandial Changes in Plasma Glucose Concentrations
Description: Incremental area under the curve (iAUC) of plasma glucose concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

6. Secondary Outcome: Postprandial Changes in Plasma Galactose Concentrations
Description: Incremental area under the curve (iAUC) of plasma galactose concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

7. Secondary Outcome: Postprandial Changes in Plasma Fructose Concentrations
Description: Incremental area under the curve (iAUC) of plasma fructose concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

8. Secondary Outcome: Postprandial Changes in Plasma VLDL-rich Triglyceride [Svedberg Flotation Rate (Sf): 20-400] Concentrations
Description: Incremental area under the curve (iAUC) of plasma VLDL-rich triglyceride [Svedberg flotation rate (Sf): 20-400] concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

9. Secondary Outcome: Postprandial Changes in Plasma Chylomicron-rich Triglyceride (Sf: >400) Concentrations
Description: Incremental area under the curve (iAUC) of plasma chylomicron-rich triglyceride (Sf: >400) concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

10. Secondary Outcome: Postprandial Changes in Plasma Lactate Concentrations
Description: Incremental area under the curve (iAUC) of plasma lactate concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

11. Secondary Outcome: Postprandial Changes in Plasma Non-esterified Fatty Acid Concentrations
Description: Incremental area under the curve (iAUC) of plasma non-esterified fatty acid concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

12. Secondary Outcome: Postprandial Changes in Plasma Beta-hydroxybutyrate Concentrations
Description: Incremental area under the curve (iAUC) of plasma beta-hydroxybutyrate concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

13. Secondary Outcome: Postprandial Changes in Plasma Uric Acid Concentrations
Description: Incremental area under the curve (iAUC) of plasma uric acid concentrations
Time Frame: 6 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Maltodextrin | Sucrose | Lactose
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT04924530/Prot_SAP_000.pdf